CLINICAL TRIAL: NCT02952313
Title: Spirox Latera™ Implant Support of Lateral Nasal Wall Cartilage (LATERAL-OR) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spirox, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-CP-301
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Latera Implant (Other): All participants have unilateral or bilateral placement of LATERA Nasal Implants.
  Interventions: Device: Nasal Implant

INTERVENTIONS:
Device: Nasal Implant

SUMMARY:
This study is being conducted to obtain outcomes data in subjects with severe to extreme class NOSE scores undergoing placement of the Spirox Latera Implant with or without concurrent septoplasty and/or turbinate reduction procedures in an operating room setting.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has Nasal Obstruction Symptom Evaluation (NOSE) Score ≥55.
2. The subject has dynamic lateral nasal wall insufficiency as confirmed by Positive Modified Cottle Maneuver22.
3. The subject is ≥18 years of age.
4. The subject is willing and able to provide informed consent and comply with the study protocol.
5. The subject is seeking treatment for nasal airway obstruction due to Nasal Valve Collapse (NVC) and is willing to undergo nasal Implant procedure alone or with septoplasty and/or a turbinate reduction procedure in an operating room setting.
6. The subject has appropriate nasal and facial anatomy to receive Latera Implant.
7. The subject agrees to follow-up examinations through twelve (12) months post operatively.
8. The subject has failed a trial of appropriate maximal medical management [e.g., nasal steroids (at least 4 weeks); antihistamines; oral decongestants; nasal strips, stents, or cones]. Failure of maximal medical management may be from lack of effectiveness or inability of subject to tolerate.

Exclusion Criteria:

1. The subject is having a concurrent Functional Endoscopic Sinus Surgery (FESS) or sinuplasty.
2. The subject has had rhinoplasty within the past twelve (12) months.
3. The subject is planning to have other concurrent rhinoplasty procedure.
4. The subject is planning to have other rhinoplasty procedures or will use external dilators within twelve (12) months after the index procedure.
5. The subject has had septoplasty and/or inferior turbinate reduction within the past six (6) months.
6. The subject has, in the view of the clinician, inappropriate fixation on their nasal airway.
7. The subject plans to have any surgical or non-surgical treatment of their nasal valve, other than the index procedure, within twelve (12) months of the study.
8. The subject has a permanent Implant or dilator in the nasal area.
9. The subject has concomitant inflammatory or infectious skin conditions or unhealed wounds in the treatment area.
10. The subject currently has active nasal vestibulitis.
11. The subject has a history of nasal vasculitis.
12. The subject is a chronic systemic steroid or recreational intra-nasal drug user.
13. The subject has had a cancerous or pre-cancerous lesion and/or has had radiation exposure in the treatment area or chemotherapy.
14. The subject has polyps or pathology other than septal deviation and/or turbinate hypertrophy and/or lateral wall insufficiency that would contribute to airway obstruction.
15. The subject has a history of a significant bleeding disorder(s) that would prevent healing of the treatment area post procedure.
16. The subject has a known or suspected allergy to poly lactic acid (PLA) or other absorbable materials.
17. The subject has a significant systemic disease such as poorly controlled diabetes which, in the investigator's opinion, could pre-dispose the subject to poor wound healing.
18. The subject is currently using nasal oxygen or continuous positive airway pressure (CPAP).
19. The subject is not a candidate for procedures conducted under general anesthesia, managed anesthesia care (MAC) or conscious sedation.
20. If female, subject is known or suspected to be pregnant or is lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Beverly Hills Aesthetic Surgical Institute, Beverly Hills, California
  - ENT Assoc. of South Florida, Boca Raton, Florida
  - The Center for Sinus, Allergy & Sleep Wellness, Boynton Beach, Florida
  - ENT of Georgia, Atlanta, Georgia
  - Chicago Nasal & Sinus Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - ENT New Orelans, Marrero, Louisiana
  - Madison ENT & Facial Plastic Surgery, New York, New York
  - Piedmont ENT, Winston-Salem, North Carolina
  - ENT & Allergy Center of Austin, Austin, Texas
  - Collin County ENT, Frisco, Texas
  - Ogden Clinic, Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stolovitzky P, Sidle DM, Ow RA, Nachlas NE, Most SP. A prospective study for treatment of nasal valve collapse due to lateral wall insufficiency: Outcomes using a bioabsorbable implant. Laryngoscope. 2018 Nov;128(11):2483-2489. doi: 10.1002/lary.27242. Epub 2018 May 14. PMID 29756407
- [Derived] Sidle DM, Stolovitzky P, O'Malley EM, Ow RA, Nachlas NE, Silvers S. Bioabsorbable Implant for Treatment of Nasal Valve Collapse with or without Concomitant Procedures. Facial Plast Surg. 2021 Oct;37(5):673-680. doi: 10.1055/s-0041-1726464. Epub 2021 Apr 14. PMID 33853139

RESULTS

PARTICIPANT FLOW:
Period: Primary Endpoint
Arm/Group | Latera Implant
Started | 113
6 Months | 106
Completed | 106
Not Completed | 7
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1
Not completed — Missed visit | 1
Period: Long-term Follow-up
Arm/Group | Latera Implant
Started (Participant with missed 6-month visit (primary endpoint) was included in later follow-up.) | 107
12-Month | 93
18-Month | 79
Completed | 75
Not Completed | 32
Not completed — Lost to Follow-up | 12
Not completed — Did not reconsent for long-term FU | 7
Not completed — Lack of Efficacy | 6
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Latera Implant: All participants have unilateral or bilateral placement of LATERA Nasal Implants.
  Nasal Implant
Arm/Group | Latera Implant
Number analyzed (Participants) | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Non-Hispanic or Latino | 102
  Ethnicity: Hispanic or Latino | 10
  Ethnicity: Unspecified | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 113
NOSE Score (100-point scale) [Mean (Standard Deviation); unit: units on a scale] — Nasal Obstruction Symptom Evaluation (NOSE) scale quantifies symptom severity of nasal obstruction. The tool is comprised of 5 questions (nasal congestion, nasal obstruction, trouble nose breathing, trouble sleeping, and difficulty breathing during exercise or exertion) that are rated from 0 (no problem) to 4 (severe problem). The scores for each item are summed, multiplied by 5, and reported on a 100-point scale. Scores of 5 to 25 indicate mild, 30-50 moderate, 55-75 severe, and 80-100 extreme symptoms.
  units on a scale | 78.5 (13.8)
NOSE Severity Classification [Count of Participants; unit: Participants]
  Severe (NOSE Scores of 55-75) | 56
  Extreme (Nose Scores of 80-100 | 57

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint is the Percent of Treatment Responders
Description: Responder is defined as a participant who has improvement of at least 1 Nasal Obstruction Symptom Evaluation (NOSE) class or at least 20% NOSE score reduction. NOSE scores. NOSE scores can range from 5 to 100, with higher scores indicating worse symptoms. Classes are mild (5-25), moderate (30-50), severe (55-75), and severe (80-100).
Time Frame: 6 months post procedure
Population: All participants with 6-month NOSE scores
Measure: Count of Participants; unit: Participants
Arm/Group | Latera Implant
Number analyzed (Participants) | 106
Participants | 101

2. Primary Outcome: Primary Safety Endpoint: Nasal Procedure and Latera™ Device-related Adverse Events
Description: Number of participants with a device-related or procedure-related adverse event
Time Frame: 6 months post procedure
Measure: Count of Participants; unit: Participants
Groups:
- Latera Implant: All participants with unilateral or bilateral placement of LATERA Nasal Implants.
Arm/Group | Latera Implant
Number analyzed (Participants) | 113
Participants | 10

3. Secondary Outcome: Percent of Treatment Responders
Description: as for outcome 1
Time Frame: 1, 3 12, 18, and 24 months post procedure.
Population: All participants with NOSE scores at the applicable visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Latera Implant
Number analyzed (Participants) | 112
Participants
  1-Month FU | 104
  3-Month FU: number analyzed (Participants) | 111
  3-Month FU | 106
  12-Month FU: number analyzed (Participants) | 93
  12-Month FU | 88
  18-Month FU: number analyzed (Participants) | 73
  18-Month FU | 70
  24-Month FU: number analyzed (Participants) | 75
  24-Month FU | 72

4. Secondary Outcome: Change in Nasal Airway Obstruction From Baseline Using the Visual Analog Scale (VAS).
Description: Change from baseline in VAS score for ability to breathe through the nose. Participants provide scores on a scale of 0 (easy to breathe through the nose) to 100 (unable to breathe through the nose). Negative values for the change from baseline indicate improvement in symptoms.
Time Frame: 1, 3, 6, 12, 18, and 24 months post procedure
Population: All participants with VAS scores at the applicable visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Latera Implant
Number analyzed (Participants) | 112
score on a scale
  1-Month FU | -40.4 [-44.4 to -36.4]
  3-Month FU: number analyzed (Participants) | 111
  3-Month FU | -46.3 [-50.3 to -42.3]
  6-Month FU: number analyzed (Participants) | 105
  6-Month FU | -45.6 [-49.7 to -41.5]
  12-Month FU: number analyzed (Participants) | 93
  12-Month FU | -47.5 [-51.9 to -43.1]
  18-Month FU: number analyzed (Participants) | 73
  18-Month FU | -48.7 [-53.6 to -43.8]
  24-Month FU: number analyzed (Participants) | 75
  24-Month FU | -51.0 [-55.9 to -46.2]

5. Secondary Outcome: Subject Satisfaction Questionnaire
Description: Participants rate whether they are satisfied or not satisfied with the procedure and cosmetic appearance after the procedure. The percent of participants reporting satisfaction with the procedure is reported.
Time Frame: 6 months
Population: All participants with satisfaction questionnaires completed at the 6-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Latera Implant
Number analyzed (Participants) | 105
Participants | 89

6. Secondary Outcome: Procedure and Device Related Adverse Events
Description: Number of participants who experience procedure or device-related adverse events.
Time Frame: After 6 months and up to 24 months post procedure
Population: All participants with follow-up beyond 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Latera Implant
Number analyzed (Participants) | 106
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events for the primary safety endpoint are reported for the 6-month period after the study procedure.
Description: Adverse events were systematically collected completion of standardized case report forms.
Arm/Group | Latera Implant
All-Cause Mortality (participants affected / at risk) | 1/113
Serious Adverse Events (participants affected / at risk) | 2/113
Other Adverse Events (participants affected / at risk) | 19/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Latera Implant (N=113)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) — Patient experienced a GI bleed 3 months after the implant procedure. Unrelated to implant or procedure.
Heart valve disease (Cardiac disorders) | 1 (1) — Pre-existing cardiac disorder with worsening symptoms requiring surgery.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Latera Implant (N=113)
Sinusitis (Infections and infestations) | 13 (16)
Implant retrieval/extrusion (Surgical and medical procedures) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Additional publications are restricted to after publication of the multicenter study results. The only other restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT02952313/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT02952313/SAP_001.pdf